CLINICAL TRIAL: NCT06749249
Title: Enjoyment Mediates Long-term Changes in Physical Activity Level in a Physical Activity on Prescription Intervention
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: Mediator study 282895
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Health Behavior; Physical Activity; Metabolic Syndrome; Primary Health Care; Adults
Keywords: Physical activity on prescription; Mediators of physical activity change
MeSH Terms: conditions — Health Behavior; Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A sufficient level of physical activity (PA) positively affects health and longevity. In Swedish healthcare, insufficiently physically active patients are offered physical activity on prescription (PAP) treatment, an individual support to increase physical activity level. This study investigates the influence of possible mediators and factors associated with a PA level change in primary care patients during a 5-year PAP intervention.

The study population includes 444 patients (56% females), aged 27 to 85 years, with metabolic risk factors and being physically inactive. The patients receive individualized PAP-treatment including PA-consultations, agreed PA recommendations with a written prescription, and structured follow-ups. Associations between 10 theoretical important mediators and factors of PA change, measured at 6 occasions, are analysed against PA level at 5 years and PA level change during the 5-year intervention.

DETAILED DESCRIPTION:
Aim:

To investigate the influence of possible mediators and factors associated with a physical activity (PA) level change in primary care patients during a 5-year physical activity on prescription (PAP) intervention.

Study design:

This is a longitudinal prospective observational cohort study with a 5-year follow-up of PAP-treatment. The treatment is carried out as part of a daily clinical primary care practice.

Study population:

The 444 patients (56% females), aged 27 to 85 years, are selected from 15 primary health care centres in Gothenburg, being physically inactive, having at least one component of the metabolic syndrome present and receiving PAP-treatment. The patients have to understand the Swedish language to fill in the questionnaires.

Intervention:

The PAP-treatment is offered by authorized personnel, educated in PA-effects and PAP-intervention and consists of an individual-based dialogue with the patient, an individually tailored recommendation of PA including a written prescription, and customized, structured support during 5 years. The patients health status, previous respectively current PA level, preferences for different physical activities, motivation, self-efficacy and readiness to change PA behavior are evaluated. An agreed individually dosed PA is written down and the support during the 5-year intervention is individually structured either by revisits or by telephone contacts.

Measurements:

The following measurements are conducted on 6 occasions during the 5-year intervention, at baseline and at the 6-month-, 1.5-, 2.5-, 3.5-, and 5-year follow-ups: PA-level, outcome expectations, enjoyment, confidence in readiness to change, self-efficacy, social support, health related quality of life, body mass index (BMI), age and sex.

Statistical analysis:

Differences between baseline and the 5-year follow-up, within the group, are analyzed using the paired sample t-test or Wilcoxon sign-rank test, based on the data level. A change score (PA at 5 year - PA at baseline) of PA is conducted, thereafter associations between theoretical important mediators of PA change (i.e., outcome expectation and confidence at baseline, and enjoyment, self-efficacy, family positive support, friends positive support and family negative support at 5 year) and PA level at 5 years and PA level change are analyzed using a linear regression. In a final step a mediation model of the mediators of PA change: enjoyment, self-efficacy, and social support and PA level at 5 years and PA level change is conducted using the lavaan package in RStudio version 1.4.1106.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive according to ACSM/AHA public health recommendation from 2007.

Having at least one component of the metS present according to the National Cholesterol Education Program (NCEP) classification.

Receiving PAP-treatment. Understanding the Swedish language.

Exclusion Criteria:

* The patient decline to participate.

Ages: 27 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included 444 patients, aged 27-85 years, with metabolic risk factors and being insufficiently physically active according to the internationally recommended minimum PA level of 150 min/week. The patients were recruited between 2010 and 2014 from 15 primary health care centres in Gothenburg, Sweden, as a convenience sample after agreeing to participate in the PAP treatment.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Change in self-reported PA-level according to the public health recommendation. | From enrollment to the end of treatment at 5 years.
  Self-assessment of PA-level according to American college of sports medicine (ACSM) and American heart association (AHA) public health recommendation 2007. The patient responds to two PA questions, where 30 minutes of moderate-intensity PA per day results in 1 point and 20 minutes of more vigorous-intensity PA per day results in 1.7 point during each specific day of the week. A value of <5 points indicates an inadequate PA level corresponding to <150 min/week at a moderate intensity level alternatively 75 min/week at a high intensity level.

SECONDARY OUTCOMES:
Outcome expectations - Outcome Expectations for Exercise-2 Scale (OEE-2) | From enrollment to the end of treatment at 5 years
  Including 13 positively- (e.g. "Helps me feel less tired"), or negatively- (e.g. "Is something I avoid because it causes me to be short of breath") worded items rated on a 5-point Likert scale (1: Strongly agree, 5: Strongly disagree). After a reverse-scoring of the positive OEE items, the numerical values for each response were summarised and divided by the number of items where a highly valued outcome expectation from the patient gave a high total score.
Enjoyment - Physical Activity Enjoyment Scale (PACES) | From enrollment to the end of treatment at 5 years.
  Including 16 positively- (e.g." I think it´s fun", "It gives me energy"), or negatively- (e.g. "I feel bored", "I don´t like it") worded items rated on a 5-point Likert scale (1: Does not apply at all, 5: Truly applies). The negative PACES items were reversed-scored, and the responses were added to a score ranging from 16 to 80 where higher scores indicated higher estimated enjoyment.
Confidence in readiness to change | From enrollment to the end of treatment at 5 years.
  Was assessed with the question "How confident are you about succeeding with changing PA level?" (36, 54) via a 100-mm visual analogue scale (VAS) anchored at each end with words that describe the minimum (Not at all) and maximum (Very) extremes.
Self-efficacy expectations - Self-Efficacy for Exercise Scale (SEE) | From enrollment to the end of treatment at 5 years.
  The patient´s self-efficacy in being able to exercise 3 times a week for 20 min despite obstacles was measured with a questionnaire including 9 items (e.g. "The weather was bothering you", "You had to exercise alone") rated on an ordinal 10-point scale (1: Not confident, 10: Very confident) where the item scores were summarised and divided by the numbers of responses.
Social support - Social support for exercise scale (SSES) | From enrollment to the end of treatment at 5 years.
  Including 13 items - 11 positively-worded (participation and involvement) and 2 negatively-worded (rewards and punishments) rated on a 5-point Likert scale (1: None, 5: Very often). The item scores were summarised in three subgroups: Family support - positive, Friend support - positive, and Family support - negative.
Health related quality of life - the Swedish version of the Short Form 36 (SF-36 Standard Swedish Version 1.0) | From enrollment to the end of treatment at 5 years.
  Includes 36 questions generating 8 health concepts that were grouped into a physical component summary (PCS) and mental component summary (MCS). The PCS and MCS are converted to 0 to 100 points, with higher values representing better HRQoL.
Body mass index - BMI | From enrollment to the end of treatment at 5 years.
  Measured body weight in kilograms (kg), with light clothing and without shoes to the nearest 0.1 kg using an electric scale (Carl Lidén AFW D300, Jönköping, Sweden) and measured body height in meters (m), measured in an upright position without shoes to the nearest 0.5 cm using a scale fixed to the wall (PEM 136, Hultafors, Sweden). Weight and height will be combined and calculated to report BMI in kg/m2.

OTHER OUTCOMES:
Socio demographic data. | From enrollment to the end of treatment at 5 years.
  Age (years), sex (female-male) were also measured.

IPD SHARING:
Plan to Share IPD: Yes
Unidentifiable patient data for all primary and secondary outcome measures will be made available in a source data file (XLSX) in published article.
Time Frame: A source data file will be available in section "Supporting information" in published article.

REFERENCES:
- [Background] Buffey AJ, Herring MP, Langley CK, Donnelly AE, Carson BP. The Acute Effects of Interrupting Prolonged Sitting Time in Adults with Standing and Light-Intensity Walking on Biomarkers of Cardiometabolic Health in Adults: A Systematic Review and Meta-analysis. Sports Med. 2022 Aug;52(8):1765-1787. doi: 10.1007/s40279-022-01649-4. Epub 2022 Feb 11. PMID 35147898
- [Background] Onerup A, Arvidsson D, Blomqvist A, Daxberg EL, Jivegard L, Jonsdottir IH, Lundqvist S, Mellen A, Persson J, Sjogren P, Svanberg T, Borjesson M. Physical activity on prescription in accordance with the Swedish model increases physical activity: a systematic review. Br J Sports Med. 2019 Mar;53(6):383-388. doi: 10.1136/bjsports-2018-099598. Epub 2018 Nov 9. PMID 30413421
- [Background] Lundqvist S, Borjesson M, Larsson MEH, Cider A, Hagberg L. Which patients benefit from physical activity on prescription (PAP)? A prospective observational analysis of factors that predict increased physical activity. BMC Public Health. 2019 May 2;19(1):482. doi: 10.1186/s12889-019-6830-1. PMID 31046720
- [Background] Lindsay Smith G, Banting L, Eime R, O'Sullivan G, van Uffelen JGZ. The association between social support and physical activity in older adults: a systematic review. Int J Behav Nutr Phys Act. 2017 Apr 27;14(1):56. doi: 10.1186/s12966-017-0509-8. PMID 28449673
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Klompstra L, Deka P, Almenar L, Pathak D, Munoz-Gomez E, Lopez-Vilella R, Marques-Sule E. Physical activity enjoyment, exercise motivation, and physical activity in patients with heart failure: A mediation analysis. Clin Rehabil. 2022 Oct;36(10):1324-1331. doi: 10.1177/02692155221103696. Epub 2022 Jun 9. PMID 35678610
- [Background] Chen Y, Jin X, Chen G, Wang R, Tian H. Dose-Response Relationship Between Physical Activity and the Morbidity and Mortality of Cardiovascular Disease Among Individuals With Diabetes: Meta-Analysis of Prospective Cohort Studies. JMIR Public Health Surveill. 2024 Aug 19;10:e54318. doi: 10.2196/54318. PMID 38780218
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] Eynon M, Foad J, Downey J, Bowmer Y, Mills H. Assessing the psychosocial factors associated with adherence to exercise referral schemes: A systematic review. Scand J Med Sci Sports. 2019 May;29(5):638-650. doi: 10.1111/sms.13403. Epub 2019 Mar 7. PMID 30742334
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Kendzierski D, DeCarlo KJ. Physical activity enjoyment scale: two validation studies. Journal of Sport & Exercise Psychology. 1991;13(1)
- [Background] Barnett I, Guell C, Ogilvie D. The experience of physical activity and the transition to retirement: a systematic review and integrative synthesis of qualitative and quantitative evidence. Int J Behav Nutr Phys Act. 2012 Aug 16;9:97. doi: 10.1186/1479-5868-9-97. PMID 22897911
- [Background] Prochaska JO. Decision making in the transtheoretical model of behavior change. Med Decis Making. 2008 Nov-Dec;28(6):845-9. doi: 10.1177/0272989X08327068. Epub 2008 Nov 17. PMID 19015286
- [Background] Resnick B. Reliability and validity of the Outcome Expectations for Exercise Scale-2. J Aging Phys Act. 2005 Oct;13(4):382-94. doi: 10.1123/japa.13.4.382. PMID 16301750
- [Background] Hagberg LA, Lindahl B, Nyberg L, Hellenius ML. Importance of enjoyment when promoting physical exercise. Scand J Med Sci Sports. 2009 Oct;19(5):740-7. doi: 10.1111/j.1600-0838.2008.00844.x. Epub 2008 Aug 5. PMID 18694433
- [Background] Baranowski T, Anderson C, Carmack C. Mediating variable framework in physical activity interventions. How are we doing? How might we do better? Am J Prev Med. 1998 Nov;15(4):266-97. doi: 10.1016/s0749-3797(98)00080-4. PMID 9838973
- [Background] Rhodes RE, Boudreau P, Josefsson KW, Ivarsson A. Mediators of physical activity behaviour change interventions among adults: a systematic review and meta-analysis. Health Psychol Rev. 2021 Jun;15(2):272-286. doi: 10.1080/17437199.2019.1706614. Epub 2020 Jan 8. PMID 31875768
- [Background] Kahlert D. Maintenance of physical activity: Do we know what we are talking about? Prev Med Rep. 2015 Mar 1;2:178-80. doi: 10.1016/j.pmedr.2015.02.013. eCollection 2015. PMID 26844069
- [Background] Lundqvist S, Cider A, Larsson MEH, Hagberg L, Bjork MP, Borjesson M. The effects of a 5-year physical activity on prescription (PAP) intervention in patients with metabolic risk factors. PLoS One. 2022 Oct 31;17(10):e0276868. doi: 10.1371/journal.pone.0276868. eCollection 2022. PMID 36315564
- [Background] Bourke E, Rawstorn J, Maddison R, Blakely T. The effects of physical inactivity on other risk factors for chronic disease: A systematic review of reviews. Prev Med Rep. 2024 Aug 22;46:102866. doi: 10.1016/j.pmedr.2024.102866. eCollection 2024 Oct. PMID 39257876
- [Background] Joseph MS, Tincopa MA, Walden P, Jackson E, Conte ML, Rubenfire M. The Impact Of Structured Exercise Programs On Metabolic Syndrome And Its Components: A Systematic Review. Diabetes Metab Syndr Obes. 2019 Nov 18;12:2395-2404. doi: 10.2147/DMSO.S211776. eCollection 2019. PMID 31819565